CLINICAL TRIAL: NCT01293019
Title: Impact of an Osteopathic Manipulative Treatment on Pain of Adult Patients With Cystic Fibrosis - a Pilot Study
Brief Title: Osteopathic Treatment in Adult Patients With Cystic Fibrosis
Acronym: MUCOSTEO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Vaincre la Mucoviscidose (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P 080701
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Cystic Fibrosis; Back Pain; Neck Pain; Chest Pain
Keywords: Complementary and alternative medicine; Osteopathic treatment
MeSH Terms: conditions — Cystic Fibrosis; Back Pain; Neck Pain; Chest Pain | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental (Experimental): Osteopathic treatment
  Interventions: Procedure: Osteopathic treatment
- Placebo (Placebo Comparator): Sham osteopathic treatment
  Interventions: Procedure: Sham Placebo
- Usual care (Active Comparator): Classic treatment of cystic fibrosis patients
  Interventions: Procedure: Usual care

INTERVENTIONS:
Procedure: Osteopathic treatment — Real treatment of osteopathy
  Other Names: Real treatment of osteopathy
  Arms: Experimental
Procedure: Sham Placebo — Sham treatment of osteopathy
  Other Names: Sham treatment of osteopathy
  Arms: Placebo
Procedure: Usual care — Classical treatment of pain in cystic fibrosis patients
  Other Names: Classical treatment of pain in cystic fibrosis patients
  Arms: Usual care

SUMMARY:
To study the contribution of osteopathy on the reduction of pain in adult patients with cystic fibrosis

DETAILED DESCRIPTION:
To compare the impact of osteopathic treatment to a placebo of osteopathic treatment and to usual care on pain at 6 months in adult patient with cystic fibrosis localized to chest, cervical, dorsal neck or back.

ELIGIBILITY:
Inclusion criteria :

* Diagnosis of cystic fibrosis ( positive sweat test and / or presence of 2 disease causing mutations in the CFTR gene
* Age > 18 years
* Patient with chronic chest , neck or back pain
* Written Informed Consent
* with health insurance

Exclusion criteria :

* regular follow-up by an osteopathic physician in the previous 3 months
* patients awaiting lung transplantation
* history of lung transplantation
* pregnancy
* understanding disorders preventing the patient to apply the study
* participation in another clinical interventional study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-11; Primary Completion 2011-04 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pain score | at 6 months

SECONDARY OUTCOMES:
quality of life scores | at 6 months
Co-interventions | at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Hubert, MD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Cochin Hospital, Paris, France

REFERENCES:
- [Derived] Hubert D, Soubeiran L, Gourmelon F, Grenet D, Serreau R, Perrodeau E, Zegarra-Parodi R, Boutron I. Impact of osteopathic treatment on pain in adult patients with cystic fibrosis--a pilot randomized controlled study. PLoS One. 2014 Jul 16;9(7):e102465. doi: 10.1371/journal.pone.0102465. eCollection 2014. PMID 25029347